CLINICAL TRIAL: NCT00207311
Title: A Multi-Centered, Prospective, Randomized, Placebo-Controlled Clinical Trial for the Treatment of Significant Steatosis or NASH With Xenical Followed by Treatment of Hepatitis C (HCV) With PEG-Interferon Alpha-2a/Copegus
Brief Title: Study for the Treatment of Significant Steatosis With Xenical Followed by Treatment of Hepatitis C With Pegasys/Copegus
Acronym: HCVNASH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: Hoffmann-La Roche (Industry); The Geneva Foundation (Other)
Responsible Party: Principal Investigator, Stephen A Harrison, Principal Investigator, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C.2004.140
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Fatty Liver; Hepatitis C
Keywords: Hepatitis C; Fatty Liver; NASH; Steatohepatitis
MeSH Terms: conditions — Fatty Liver; Hepatitis C | interventions — Orlistat; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Xenical placebo (Placebo Comparator): Xenical placebo PO three times daily with meals plus enrollment into the Xenicare program for 36 weeks followed by 48 weeks of therapy with Pegasys (180mcg/ml) plus weight based ribavirin for HCV genotype 1 or 4 and 24 weeks of therapy with Pegasys (180mcg/ml) plus 800mg ribavirin for HCV genotypes 2 and 3.
  Interventions: Behavioral: Xenicare Program
- Xenical (orlistat) (Active Comparator): Xenical (orlistat) 120mg PO three times daily with meals plus enrollment into the Xenicare program for 36 weeks followed by 48 weeks of therapy with Pegasys (180mcg/ml) plus weight based ribavirin for HCV genotype 1 or 4 and 24 weeks of therapy with Pegasys (180mcg/ml) plus 800mg ribavirin for HCV genotypes 2 and 3.
  Interventions: Drug: Xenical, Pegasys, Copegus

INTERVENTIONS:
Drug: Xenical, Pegasys, Copegus — Xenical 120mg three times daily for 36 weeks or xenical placebo (Arm 1). Pegasys 180 mcg weekly for 48 weeks. Ribavirin daily for 48 weeks.
  Other Names: Xenical (orlistat); Pegasys (PEG-Interferon alpha-2a)
  Arms: Xenical (orlistat)
Behavioral: Xenicare Program — Xenicare program for 36 weeks.
  Other Names: Xenical placebo; Pegasys (Peg interferon alpha-2a)
  Arms: Xenical placebo

SUMMARY:
This is a prospective, multi-center, randomized, placebo-controlled trial in subjects with histological evidence of > 33% hepatic steatosis or nonalcoholic steatohepatitis (NASH) and chronic hepatitis C. Patients who have not been previously treated for hepatitis C (treatment naive) will be enrolled.

DETAILED DESCRIPTION:
Recent evidence suggests that patients with concomitant chronic HCV infection and NASH or significant hepatic steatosis (>33%) respond less well to standard antiviral therapy. As previously noted, up to 10% of patients with chronic HCV infection will have concomitant NASH and an even greater percentage will have associated hepatic steatosis. No prospective studies to date have evaluated the sustained viral response rates to standard antiviral therapy in this group of patients who were previously treated with a medication to eliminate or improve the underlying NASH and/or hepatic steatosis.

Primary Outcome: To determine if decreasing the amount of NASH or hepatic steatosis in overweight (BMI >27 kg/m2) HCV patients results in improved overall SVR to PEGASYS and Copegus.

Secondary Outcome: 1.To determine the amount of steatosis, necroinflammatory activity, and fibrosis change in a group of participants with chronic hepatitis C and NASH or significant steatosis treated with Xenical vs. placebo for 36 weeks. 2. To assess for a difference in insulin resistance, as measured by the QUICKI score, before and after treatment with Xenical or Xenical placebo and diet and exercise.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be willing to give written informed consent and be able to adhere to dose and visit schedules.
* HCV-Ab or HCV-RNA by PCR Positive for at least 6 months
* Serum positive for HCV-RNA by PCR assay
* Treatment naïve participants who have hepatitis C with genotype 1, 2, 3, or 4
* Body mass index >27
* Liver biopsy within 12 months with a pathology report confirming the histological diagnosis consistent with CHCand NASH or hepatic steatosis of >33%
* Compensated liver disease with minimum hematological, biochemical, and serologic criteria at the Enrollment Visit (WNL = within normal limits):

  * Hemoglobin values of <12 gm/dL for females and <13 gm/dL for males
  * WBC <3,000/ mm3
  * Neutrophil count < 1,500/mm3
  * Platelets <65,000/ mm3
  * Direct bilirubin within 20% of ULN
  * Indirect bilirubin WNL
  * Albumin > 3 gm/dL
  * creatinine < 20% of ULN
  * TSH WNL
  * Alpha fetoprotein value < 100 ng/mL
* Reconfirmation and documentation that sexually active female subjects of childbearing potential are practicing adequate contraception method, or monogamous relationship with a male partner who has had a vasectomy or is using a condom + spermicide) during the treatment period and for six months following the last dose of study medication
* Reconfirmation that sexually active male subjects are practicing two acceptable methods of contraception

Exclusion Criteria:

* Women who are pregnant or breast-feeding
* Males whose female partner is pregnant
* No other Thiazolidinedione after liver biopsy and/or during the entire study
* Hepatitis C of non-genotype 1,2,3 or 4
* Previous anti-viral therapy for treatment of Hepatitis C
* Suspected hypersensitivity to interferon, PEG-interferon, ribavirin, Xenical
* Any other cause for liver disease other than chronic hepatitis C and NASH or steatosis, including but not limited to:

  * Hemochromatosis
  * Alpha-1 antitrypsin deficiency
  * Co-infection with HBV
  * Wilson's disease
  * Autoimmune hepatitis
  * Alcoholic liver disease
  * Drug-related liver disease
* Any condition that would prevent the subject from having a liver biopsy
* Hemoglobinopathies (e.g., Beta Thalassemia)
* Evidence of advanced liver disease
* Patients with organ transplants other than cornea and hair transplant
* Any known preexisting medical condition that could interfere with the subject's participation in and completion of the protocol such as:

  * Preexisting psychiatric condition, especially severe depression, or a history of severe psychiatric disorder, such as major psychoses, suicidal ideation and/or suicidal attempt are excluded
  * CNS trauma or preexisting/active seizure disorders uncontrolled with medication
  * Significant cardiovascular dysfunction within the past 12 months
  * Poorly controlled diabetes mellitus
  * Chronic pulmonary disease with documented pulmonary hypertension
  * Immunologically mediated disease (Crohn's disease, ulcerative colitis), rheumatoid arthritis, idiopathic thrombocytopenia purpura, systemic lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis, clinical cryoglobulinemia with vasculitis
* Any medical condition requiring, or likely to require chronic systemic administration of steroids
* Evidence of an active or suspected cancer or a history of malignancy where the risk of reoccurrence is ≥ 20% within 2 years
* Active clinical gout
* Substance abuse
* Participants not willing to be counseled/abstain from alcohol
* Participants with clinically severe retinal abnormalities
* Any other condition that in the opinion of the investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in and completing the protocol
* Known positive HIV
* Inability/unwillingness to provide informed consent or abide by the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Sustained virological response (SVR) defined as the percentage of participants with undetectable HCV-RNA as measured by the Roche AMPLICORTM HCV Test, v 2.0 (detection limit 50 IU/mL) at 24 weeks post completion of the treatment period | 110 weeks

SECONDARY OUTCOMES:
Hepatic steatosis, necroinflammatory activity and fibrosis improvement at week 36 as determined by Dr. Elizabeth Brunt at Saint Louis University | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A Harrison, MD, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States